CLINICAL TRIAL: NCT02807324
Title: Women Specific Cardiac Recovery After Preeclampsia
Acronym: WeCare
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL52556.068.15; Local Ethical Commission (Other: METC 152019)
Record Dates: First submitted 2016-06-08; First posted 2016-06-21 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Pre-Eclampsia; Pregnancy; HELLP Syndrome; Intrauterine Growth Restriction
MeSH Terms: conditions — Pre-Eclampsia; HELLP Syndrome; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for microRNA analyses
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Controls: Controls are women (18 years or older) with an uncomplicated pregnancy (i.e no foetal or maternal placental complications, such as pregnancy induced hypertension, preeclampsia or HELLP-syndrome, or small for gestational birth infancies)
  Interventions: Other: Venapunction
- Early PE with IUGR: These cases consist of women (18 years or older) with preeclampsia (PE) and/or HELLP syndrome in the current pregnancy (PE is defined as hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg) developed after 20 weeks of pregnancy with de novo proteinuria (≥ 300 mg/ 24 hours)) Cases will be subdivides in early and late PE, with or without IUGR (Early PE is defined as the occurence of PE < 34 weeks of gestation, whereas late PE is defined as the occurence of PE ≥ 34 weeks of gestation. IUGR is defined as birthweight below the 10th percentile).
  Interventions: Other: Venapunction
- Early PE without IUGR: Cases consist of women (18 years or older) with preeclampsia (PE) and/or HELLP syndrome in the current pregnancy (PE is defined as hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg) developed after 20 weeks of pregnancy with de novo proteinuria (≥ 300 mg/ 24 hours)) Cases will be subdivides in early and late PE, with or without IUGR (Early PE is defined as the occurence of PE < 34 weeks of gestation, whereas late PE is defined as the occurence of PE ≥ 34 weeks of gestation. IUGR is defined as birthweight below the 10th percentile).
  Interventions: Other: Venapunction
- Late PE with IUGR: Cases consist of women (18 years or older) with preeclampsia (PE) and/or HELLP syndrome in the current pregnancy (PE is defined as hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg) developed after 20 weeks of pregnancy with de novo proteinuria (≥ 300 mg/ 24 hours)) Cases will be subdivides in early and late PE, with or without IUGR (Early PE is defined as the occurence of PE < 34 weeks of gestation, whereas late PE is defined as the occurence of PE ≥ 34 weeks of gestation. IUGR is defined as birthweight below the 10th percentile).
  Interventions: Other: Venapunction
- Late PE without IUGR: Cases consist of women (18 years or older) with preeclampsia (PE) and/or HELLP syndrome in the current pregnancy (PE is defined as hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg) developed after 20 weeks of pregnancy with de novo proteinuria (≥ 300 mg/ 24 hours)) Cases will be subdivides in early and late PE, with or without IUGR (Early PE is defined as the occurence of PE < 34 weeks of gestation, whereas late PE is defined as the occurence of PE ≥ 34 weeks of gestation. IUGR is defined as birthweight below the 10th percentile).
  Interventions: Other: Venapunction
- HELLP syndrome: Cases consist of women (18 years or older) with HELLP syndrome in the current pregnancy (defined as (1) the presence of microangiopathic hemolytic anemia with abnormal blood smear, low serum haptoglobin and elevated lactate dehydrogenase (LDH) levels, (2) aspartate transaminase (ASAT) above 70 IU/L and lactate dehydrogenase (LD) above 600 IU/L or bilirubin more than 1.2 mg/dL, (3) platelet count below 100 x 10^9 L-1 )
  Interventions: Other: Venapunction

INTERVENTIONS:
Other: Venapunction — The only invasive procedure is a venapunction where 75 ml blood will be extracted. The only unfavourable side effect can be a small hematoma (rare).

SUMMARY:
Pregnancy is considered a cardiovascular (CV) stress test, and complicated pregnancies are associated with an increased risk for cardiovascular disease (CVD) later in life. Moreover, it is known that often the pregnancy induced CV adaptation does not resolve completely after a short postpartum (PP) period and it is not clear whether these induced changes will resolve over a longer period of time (i.e. in the upcoming months/years after delivery). Understanding the cardiac adaptation during pregnancy and the reversal process in the postpartum period, as well as the factors that influence this these processes, may provide us not only insight in this mechanism, but may help us in identifying factors that may be target points for modification.

DETAILED DESCRIPTION:
The main goal of this study is to explore the pattern of physiologic and pathophysiologic cardiac recovery after a preeclamptic pregnancy compared to a normotensive pregnancy, up till 18 months PP.

This study is a longitudinal cohort study. The first measurement will be performed upon admittance for induction of labour or caesarean section, which corresponds with 48-24 hours before delivery. Further measurements will be performed in clusters at PP intervals of: 24-48 hours, 3 weeks, 6 weeks, 3 months, 6 months, 12 months and 18 months. Cases will also receive an additional baseline measurement upon PE diagnosis.

Cases consist of women with preeclampsia (PE) and/or HELLP syndrome in the current pregnancy (early and late PE, with or without intra uterine growth restriction (IUGR)), whereas controls are women with an uncomplicated pregnancy. 290 women in total will be included. Inclusion will of case subjects will occur upon diagnosis, inclusion of controls will occur before delivery.

The first visit of this study will be performed upon admittance after PE diagnosis for cases, and for controls while the participant is administered for the induction of labour or caesarean section, thus an extra visit is not necessary. This is also true for the first postpartum (PP) measurements. The next 6 visits will be after the participant is discharged from the hospital and extra visits are necessary, except for the 6 weeks PP visit, which is a routine visit. The frequent visits may cause some discomfort, especially since our participants are young mothers who still need to take care of their child. During the measurement, one of our co-workers will assist in taking care of the newborn if necessary, so that the participant can bring her child with her. Each of the visits will last approximately 2 hours in the MUMC+. The only invasive procedure is a venapunction where 75 ml blood will be extracted. The only unfavourable side effect can be a small hematoma (rare). Clinically, participants will be advised based on their risk profile following standard "cardiovascular (CV) risk management". Transthoracic echocardiography, glycocalyx measurements and a FibroScan will be performed. Experience shows that this investigation is not experienced as uncomfortable. Also, 3 liters of exhaled air will be collected for VOCs analysis. All measurements will be performed or supervised by an experienced researcher. These investigations are already approved previously in other METC applications (CMO-nr: 2008/226; 2009/004; 10-2-066). The other measurements (questionnaires, blood pressure (BP), weight measurement, urine collection, glycocalyx measurement, FibroScan and exhaled air collection) do not cause any discomfort for the patient besides the time that it takes. On the other hand, potential health improvement and early detection of CV risk profiles and initiation of already existing effective prevention strategies that improve lifestyle are important benefits.

For potential participants who find the number of extra visits too great a burden, a short track version of the study is available with less postpartum visits. the first 3 measurement moments do not differ between both versions. However, after the first PP measurement, 24-48hrs after delivery, they will only have one more additional visit at 12 months PP, but we will include a coronary CTA, an MFD and carotid IMT measurement.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years
* Controls: Women with an uncomplicated pregnancy at the moment of inclusion (i.e no foetal or maternal placental complications, such as pregnancy induced hypertension, preeclampsia or HELLP-syndrome, or small for gestational birth infancies)
* Cases: Women diagnosed with a preeclamptic pregnancy at the moment of inclusion

Exclusion Criteria:

* Women with an auto-immune disease prior to the complicated pregnancy
* Chronic hypertension prior to the complicated pregnancy
* Renal disease prior to the complicated pregnancy
* Women who do not want to be informed about the results of the tests, or women who do not want their general practitioner and specialist(s) to be informed about the test results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Controls will be recruited at the outpatient clinic if a planned induction or C-section is indicated due to any obstetric reason other than placental insufficiency or pregnancy related hypertensive disease. Cases will be recruited at the MUMC+, since the current guideline in the Netherlands states that women diagnosed with preeclampsia should be referred to specialist care in the hospital.
Sampling Method: Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2016-06; Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The pattern of cardiac recovery | 4 years
  The pattern of cardiac recovery in terms of cardiac geometry (measured by relative wall thickness, left ventricular mass and cardiac dimension such as LV end systolic and diastolic diameters, atrial diameters etc..), systolic and diastolic function (measured by ejection fraction (EF%) and E/A ratio) and miRNA expression after a preeclamptic pregnancy compared to a normotensive pregnancy

SECONDARY OUTCOMES:
The prevalence of abnormal cardiac findings | 4 years
  The prevalence of abnormal cardiac findings amongst participants, such as, Concentric remodeling (based on relative wall thickness (RWT) and LVmass (gr/m2)), left ventricular (LV) hypertrophy (based on LVmass (gr/m2)), LV segmental myocardial impaired relaxation, LV segmental myocardial impaired contractility, Global systolic and diastolic dysfunction (based on ejection fraction (%) and E/A ratio respectively).
Overall health and lifestyle - Metabolic syndrome | 4 years
  The number of participants with metabolic syndrome (MetS). The MetS is a cluster of risk factors which consists of cardio-metabolic abnormalities (insulin resistance and/or impaired glucose tolerance, low high density lipoprotein (HDL) cholesterol, high triglycerides (TG)) and cardiovascular mechanical stress indicators (elevated BP, micro albuminuria, obesity). We will define the MetS based on The World Health Organisation (WHO) criteria. It consists of impaired glucose regulation, diabetes mellitus or insulin resistance with at least two of the following criteria: Elevated TG (≥1.7 nmol/l) or reduced HDL-cholesterol (< 1.0 mmol/l),Elevated BP (≥140/85mmHg), Central obesity (waist-hip ratio > 0.85 or BMI > 30 kg/m2), Micro-albuminuria (> 0.30 g/mmol creatinine)
Overall health and lifestyle - Questionnaires | 4 years
  The prevalence of cardiovascular risk factors amongst participants (determined via questionnaires).The questionnaires contains questions about daily exercise, eating and drinking habits (mainly the consumption of fruits and vegetables), and smoking/alcohol/drugs consumption. Lifestyle is known to affect the risk for CVD.By exploring lifestyle factors in both subjects and controls, we will be able to determine the (confounding) contributio of lifestyle factors for the increased risk of CVD after PE. Consequently, we will be able to study the contribution of PE independent of lifestyle on the development of CVD.
Overall health and lifestyle - Microcirculation | 4 years
  The number of participants with an increased perfused boundary region (PBR), as measures with Glycocheck. The main read-out parameter of the glycocheck machine is the perfused boundary region (PBR). In short, the endothelial glycocalyx constitutes a protective barrier for the vessel wall, which limits the proximity of erythrocytes to the endothelial cells in the microvasculature, causing the PBR to be small in healthy conditions. In contrast, perturbation of the glycocalyx allows deeper cell penetration into the glycocalyx, leading to an increase in PBR. Monitoring of the PBR, therefore, gives information about the barrier properties of the glycocalyx and the state of the microvascular system.
Overall health and lifestyle - Kidney function | 4 years
  The number of participants with a decreased kidney function, measured by abnormal lab values of a urine sample, such as total protein, creatinine and micro-albumin.
VOCs analysis | 4 years
  The highest discriminative pattern of VOCs (Volatile Oxidized Compounds) between PE patients, HELLP syndrome patients, PE + HELLP syndrome patients and healthy control pregnancies.
FibroScan | 4 years
  Differences in metabolism, liver stiffness, fibrosis and steatosis of the liver between PE patients, HELLP syndrome patients, PE + HELLP syndrome patients and healthy control pregnancies at the time of diagnosis and over time.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Spaanderman, MD, PhD, Principal Investigator — Maastricht University Medical Center (MUMC+)
Locations (1):
- Maastricht University Medical Center (MUMC+), Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No